CLINICAL TRIAL: NCT00877110
Title: Phase I Study of Anti-GD2 3F8 Antibody and Allogeneic Natural Killer Cells for High-Risk Neuroblastoma
Brief Title: Anti-GD2 3F8 Antibody and Allogeneic Natural Killer Cells for High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-011; MSKCC09011 FDR004128 (Other Grant/Funding Number: FDR004128)
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Neuroblastoma; Bone Marrow, Sympathetic Nervous System
Keywords: BETA-D-GLUCAN; CYCLOPHOSPHAMIDE (CYTOXAN); MAB 131 I - 3F8; TOPOTECAN; VINCRISTINE; Neuroblastoma; 09-011
MeSH Terms: conditions — Neuroblastoma | interventions — Cyclophosphamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy, allogeneic NK cells, 3F8 (Experimental): This is a phase I study to assess the safety and feasibility of combining HLA-mismatched (KIR ligand incompatible) NK cells with 3F8 in high-risk NB patients. Following chemotherapy, patients will be treated in sequential groups of 3 patients/dose of NK cells. Four dose levels of NK cells, starting at dose level I, will be evaluated in this treatment protocol. In the unlikely case toxicity is encountered at dose level I, patients will then be treated at the lower dose level 0. Patients can receive up to 3 cycles of treatment on protocol. For subsequent cycles, patients will be treated at either less than or at the same dose level of NK cells as their first cycle.
  Interventions: Drug: cyclophosphamide, vincristine, topotecan ,allogeneic NK cells & 3F8

INTERVENTIONS:
Drug: cyclophosphamide, vincristine, topotecan ,allogeneic NK cells & 3F8 — Patients will receive combination chemotherapy with intravenous (IV) cyclophosphamide 70mg/kg/day (for patients with body weight<70kg) or 2100mg/m2/day (for patients with body weight ≥70kg) for two days, IV vincristine 0.067mg/kg or 2mg/m2/day (lower of the two doses to be chosen; maximum 2mg) for one day, and IV topotecan 2.4 mg/m2/day for 3 days during their first cycle. If receiving a second and/or third cycle, the only chemotherapy patients will receive is cyclophosphamide at 50 mg/kg/day for 2 days. On Day 0, patients will receive a single dose of allogeneic NK cells isolated from a HLA-haploidentical related donor. On day +3, the patient will start daily infusion of 3F8 for 5 days. The treatment schedule may require minor adjustment by ±1 day as clinically indicated (e.g. due to PDH closure for holidays or due to inclement weather).

SUMMARY:
Funding Source - FDA OOPD FDR004128

The goal of this study is to see if it is safe and feasible to give chemotherapy, natural killer (NK) cells, and an antibody called 3F8. The NK cells must come from a family member who shares half of the HLA proteins which are immune proteins important in transplant. NK cells are a type of white blood cell. They can recognize and kill abnormal cells in the body and can work together with antibodies to kill target cells. The antibody 3F8 specifically recognizes a protein present on the target cancer cell.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria, i.e., histopathology (confirmed by the MSKCC Department of Pathology) or bone marrow metastases plus high urine catecholamine levels
* High-risk NB as defined by risk-related treatment guidelines and the International NB Staging System,57 i.e., stage 4 with (any age) or without (>365 days of age) MYCN amplification, MYCN-amplified stage 3 (unresectable; any age), or MYCN-amplified stage 4S.
* Patients must have a history of tumor progression or persistent disease or failure to achieve complete response following standard therapy.
* Patients must have evaluable (microscopic marrow metastasis, elevated tumor markers, positive MIBG or PET scans) or measurable (CT, MRI) disease documented after completion of prior systemic therapy.
* Disease staging approximately within one month of treatment.
* Human anti-mouse antibody (HAMA) titer <1000 Elisa units/ml if applicable
* Available autologous stem cells: ≥2 x 106 CD34+ cells/kg
* Adequate cardiac function as measured by echocardiogram
* Eligible NK donor
* Signed informed consent indicating awareness of the investigational nature of this program.

Donor Eligibility

* Donor is blood-related and HLA-haploidentical to the recipient.
* Donor has undergone serologic testing for transmissible diseases as per blood banking guidelines for organ and tissue donors. Tests include but are not limited to: HepBsAg, HepBsAb, HepBcAb, HepC antibody, HIV, HTLV I and II, VZV, CMV and VDRL, West Nile Virus and Chagas screen. Donor must have normal negative test results for HIV, HTLV I and II, and West Nile Virus. Donor exposure to other viral pathogens will be discussed on a case-by-case basis by the investigators.
* Donor must be able to undergo leukopheresis for total volume of 10-15 liters.
* There is no age restriction for the donor.

Exclusion Criteria:

* Patients with CR/VGPR disease
* Existing severe major organ dysfunction, i.e., renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity > or = to grade 3 except for hearing loss, alopecia, anorexia, nausea, hyperbilirubinemia and hypomagnesemia from TPN, which may be grade 3
* ANC should be >500/uL; platelet count >25K/uL.
* History of allergy to mouse proteins
* Active life-threatening infection
* HAMA titer >1000 Elisa units/ml
* Inability to comply with protocol requirements

Donor Exclusion Criteria

* Cardiac risk factors precluding ability to undergo leukopheresis
* Concurrent malignancy or autoimmune disease
* Donor is pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-04-02 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility and safety of administering allogeneic haploidentical NK infusions with 3F8 in patients with high-risk NB | 3 years

SECONDARY OUTCOMES:
Estimate the anti-NB effect of allogeneic NK infusions plus 3F8 | 3 years
Assess the impact of KIR/HLA immunogenetics on disease response to NK/3F8 | 3 years
Assess the relationship between CD16 polymorphism and ADCC in vitro | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org